CLINICAL TRIAL: NCT03870503
Title: Carbetocin Versus Oxytocin Plus Sublingual Misoprostol in the Management of Atonic Post-partum Hemorrhage (PPH) After Vaginal Delivery: a Randomized Controlled Trial
Brief Title: Carbetocin Versus Oxytocin Plus Sublingual Misoprostol in the Management of Atonic Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu/201/19
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum Hemorrhage; vaginal delivery; carbetocin; misoprostol; oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Misoprostol; carbetocin

STUDY DESIGN:
Intervention Model Description: This study will be a prospective double-blind randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be a prospective double-blind randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oxytocin (Active Comparator): The patient will be received oxytocin 20 IU by intravenous infusion
  Interventions: Drug: oxytocin
- oxytocin plus misoprostol (Active Comparator): The patient will be received oxytocin 20 IU by intravenous infusion plus 400 mc sublingual misoprostol
  Interventions: Drug: oxytocin; Drug: oxytocin plus misoprostol
- Carbetocin (Active Comparator): The patient will be received Carbetocin 100 mic gm IV
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: oxytocin — The patient will be received oxytocin 20 IU by intravenous infusion
  Other Names: Active comparator
  Arms: oxytocin; oxytocin plus misoprostol
Drug: oxytocin plus misoprostol — The patient will be received oxytocin 20 IU by intravenous infusion plus 400 mic gm sublingual misoprostol
  Other Names: Active Comparator
  Arms: oxytocin plus misoprostol
Drug: Carbetocin — The patient received Carbetocin 100 mic gm
  Other Names: Active Comparator
  Arms: Carbetocin

SUMMARY:
The objective of this study is to compare the effectiveness and safety of carbetocin vs. oxytocin plus sublingual misoprostol in the management of atonic postpartum hemorrhage (PPH)after vaginal delivery.

DETAILED DESCRIPTION:
The first cause of hemorrhage at the time of delivery is uterine atony; therefore, there is general agreement that active management of the third stage of labor is recommended.

Oxytocin is the most widely used uterotonic agent but has a half-life of only 4-10 min, that is why it is better administered as a continuous intravenous infusion to achieve sustained uterotonic activity. Carbetocin is a synthetic long-acting oxytocin agonistic analog with prolonged half-life prolonging its pharmacological effects. Its prolonged uterine activity may theoretically offer advantages over oxytocin in the management of the third stage of labor. The side-effect profile of carbetocin was not found to be different from that of Oxytocin but may prove to be advantageous when compared to Syntometrine.

ELIGIBILITY:
Inclusion Criteria:

* All participants had PPH defined as vaginal bleeding>500 ml after vaginal delivery and uterine atony confirmed by abdominal palpation

Exclusion Criteria:

* gestational age<37 weeks,
* genital tract trauma,
* coagulation defect,
* women with hypertension, preeclampsia, cardiac, renal or liver diseases, epilepsy
* known hypersensitivity to carbetocin or oxytocin.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All participants had PPH defined as vaginal bleeding>500 ml after vaginal delivery and uterine atony confirmed by abdominal palpation
Enrollment: 135 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The amount of blood loss | 6 hours post delivery
  calculation of the amount of blood loss by weighing the swabs and using pictorial charts

SECONDARY OUTCOMES:
The number of patients develop blood loss more than 1000 ml | 24 hours post delivery
  Calculation of the number of patients develop blood loss more than 1000 ml
The number of patient need blood transfusion | 24 hours post delivery
  Calculation of number of patient need blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: hany f allam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518